CLINICAL TRIAL: NCT01380184
Title: A Study to Assess the Pharmacokinetics of Ridaforolimus in Chinese Patients
Brief Title: Pharmacokinetics of Ridaforolimus (MK-8669) in Chinese Participants (MK-8669-059)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-059; MK-8669-059 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-01

CONDITIONS: Cancer, Advanced
Keywords: Relapsed cancer
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ridaforolimus 40 mg (Experimental): In Part 1 (Days 1-19), participants received ridaforolimus (MK-8669) 40 mg via oral enteric-coated tablet on Day 1; followed by no study treatment on Days 2-7; followed by two weekly sequences (Days 8-19) consisting of 5 consecutive days of ridaforolimus 40 mg and 2 consecutive days off study treatment. Following Part 1, participants underwent at least a 2-day study treatment washout prior to starting Part 2. In Part 2, participants received a weekly treatment regimen consisting of 5 consecutive days (Days 1-5) of ridaforolimus 40 mg via oral enteric-coated tablet and 2 consecutive days (Days 6-7) off study treatment. This weekly treatment regimen was repeated every subsequent week for the remainder of participation in Part 2.
  Interventions: Drug: ridaforolimus

INTERVENTIONS:
Drug: ridaforolimus — 4 enteric-coated tablets, each containing 10 mg ridaforolimus, orally (total daily dose: 40 mg)
  Other Names: MK-8669; AP23573; ridaforolimus was also known as deforolimus until May 2009

SUMMARY:
Part 1 of the study will assess the pharmacokinetics, safety, and tolerability of ridaforolimus (MK-8669) after administration of single and multiple 40 mg doses in Chinese participants with advanced cancer. Part 2 of the study is optional; participants can continue to receive the study treatment in a weekly regimen of daily oral doses of ridaforolimus 40 mg for five consecutive days followed by two days off-treatment.

ELIGIBILITY:
Inclusion criteria:

* Chinese descent with all 4 biological grandparents born in China and of Chinese descent.
* Histologically- or cytologically-confirmed metastatic or locally advanced solid tumor or lymphoma that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist.
* Performance status of ≤1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Female participants must be post-menopausal.
* Male participants must agree to use a medically-acceptable method of contraception/barrier protection during the study and for 30 days after the last dose of study treatment.
* Participants must be healthy enough to receive the study treatments (that is, meet certain laboratory value parameters).
* Life expectancy of >3 months.

Exclusion criteria:

* Chemotherapy, radiotherapy, or biological therapy within 4 weeks (6 weeks for nitrosoureas, mitomycin C, and monoclonal antibodies) prior to first dose of study treatment (Part 1/Day 1) or has not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Any other concurrent anti-cancer therapy (except luteinizing hormone releasing hormone [LHRH] analogs for prostate cancer).
* Concurrent treatment with immunosuppressive agents, including corticosteroids, at doses greater than those used for replacement therapy.
* Clinically significant abnormality on electrocardiogram (ECG) performed at the screening visit and/or prior to administration of the initial dose of study treatment.
* New York Heart Association (NYHA) Class III or IV congestive heart failure or any other significant history of cardiac disease including: myocardial infarction within the last 6 months; ventricular arrhythmia or acute congestive heart failure within the last 3 months; uncontrolled angina; or uncontrolled hypertension.
* Current participation or participation in a study with an investigational compound or device within 30 days prior to the first dose of study treatment.
* Primary central nervous system tumor, active brain metastases or leptomeningeal carcinomatosis.
* Regular use (including use of any illicit drugs or had a recent history within the last year) of drugs, or alcohol abuse.
* Pregnant or breastfeeding, or expecting to conceive within the projected duration of the study.
* Human Immunodeficiency Virus (HIV)-positive.
* Newly diagnosed (within 3 months before the first dose of study drug) or poorly controlled Type 1 or 2 diabetes.
* Required treatment with medications that are inducers or inhibitors of cytochrome P450 (CYP3A).
* Active infection or use of intravenous (IV) antibiotics, antiviral, or antifungal agents within 2 weeks prior to the first dose of the study treatment.
* Use of or intention to use herbal teas or herbal remedies (including traditional Chinese medicine, St.John's Wort, shark cartilage, etc.) from 2 weeks prior to the first dose and throughout the study.
* Anticipation of need for immunologic therapy, radiation therapy, surgery, or chemotherapy during the study.
* Past high-dose chemotherapy with stem cell rescue.
* Blood transfusion within one week of study entry.
* Inability to swallow capsules and/or documented surgical or anatomical condition that will preclude swallowing and absorbing oral medications on an ongoing basis.
* Known hypersensitivity to the components of the study treatment or its analogs or antibiotics (e.g. clarithromycin, erythromycin, azithromycin).
* Intention to consume grapefruit or grapefruit juice for approximately 2 weeks prior to first dosing until the completion of the study.
* Inadequate recovery from any prior surgical procedure or any major surgical procedure within 4 weeks prior to the first dose of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07-05 (Actual); Primary Completion 2011-10-20 (Actual); Study Completion 2012-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Liu L, Zhang W, Li W, Lv F, Xia Z, Zhang S, Liu W, Zandvliet AS, Waajen S, Zhang LX, Yan L, Li J. A phase I study of ridaforolimus in adult Chinese patients with advanced solid tumors. J Hematol Oncol. 2013 Jul 8;6:48. doi: 10.1186/1756-8722-6-48. PMID 23829943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen (15) Chinese participants with treatment-refractory advanced or relapsed cancers were enrolled in this study.
Period: Part 1 (19 Days)
Arm/Group | Ridaforolimus 40 mg
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1
Period: Washout Period (≥2 Days)
Arm/Group | Ridaforolimus 40 mg
Started | 14
Completed | 14
Not Completed | 0
Period: Part 2
Arm/Group | Ridaforolimus 40 mg
Started | 14
Completed | 0
Not Completed | 14
Not completed — Adverse Event | 5
Not completed — Disease Progression | 8
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ridaforolimus 40 mg
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  China | 15

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Experiencing Clinical and Laboratory Adverse Events (AEs)
Description: A laboratory AE (LAE) is defined as any unfavorable & unintended change in the chemistry of the body temporally associated with the use of study product, whether or not considered related to the use of the product. A clinical AE (CAE) is defined similarly but also includes changes in structure or function of the body. Serious AEs (SAEs) are those that result in one or more of the pre-specified outcome(s) that meet the criteria of seriousness, including death, life-threatening, significant disability, or hospitalization, etc. Drug-relatedness was determined by the investigator based on clinical judgement.
Time Frame: From first dose up to 30 days after last dose (Up to 26 weeks)
Population: The Safety Population consisted of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ridaforolimus 40 mg
Number analyzed (Participants) | 15
Participants
  Clinical & Laboratory AEs | 15
  Drug-related AEs | 15
  Serious AEs (SAEs) | 4

2. Primary Outcome: Lag Time (Tlag) of Ridaforolimus: Day 1
Description: Tlag is the time taken for ridaforolimus to appear in systemic circulation following oral administration. The median and full range (minimum, maximum) for Tlag after a single dose of ridafolorlimus are presented.
Time Frame: Cycle 1 Day 1: Predose and at various time points up to 24 hours postdose on Day 1; Cycle 1 is 19 days
Population: The Pharmacokinetic Evaluable population consisted of all participants who complied with the protocol sufficiently to ensure that these data will likely exhibit the effects of treatment according to the underlying scientific model and who had blood samples with concentrations above the lower limit of quantitation.
Measure: Median (Full Range); unit: Hours
Arm/Group | Ridaforolimus 40 mg
Number analyzed (Participants) | 15
Hours | 2.00 [0.97 to 8.07]

3. Primary Outcome: Area Under the Curve From 0 to Infinity (AUC0-∞) of Ridaforolimus: Cycle 1 (Cycle 1 is 19 Days)
Description: AUC0-∞ represents the total exposure to ridaforolimus and its average blood concentration multiplied by the total amount of time (extrapolated to infinity) that ridaforolimus was in the body. The (geometric) mean was calculated based on the back-transformed least-squares mean and the 95% confidence interval was determined from a linear mixed-effect model, containing a fixed effect for day and a random effect for participant, performed on natural log-transformed values. The geometric mean and back-transformed 95% confidence interval are presented for AUC0-∞.
Time Frame: Cycle 1: Predose on Day 1 and at various time points through to 24 hours postdose on Day 19; Cycle 1 is 19 days
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Ridaforolimus 40 mg
Number analyzed (Participants) | 13
ng*hr/mL | 3648 [3044 to 4372]

4. Primary Outcome: Area Under the Curve From 0 to 24 Hours (AUC0-24hr) of Ridaforolimus: Day 1, Day 19
Description: AUC0-24hr represents the total exposure to ridaforolimus and its average blood concentration multiplied by the total amount of time (extrapolated to 24 hours) that ridaforolimus was in the body. The (geometric) mean was calculated based on the back-transformed least-squares mean and the 95% confidence interval was determined from a linear mixed-effect model, containing a fixed effect for day and a random effect for participant, performed on natural log-transformed values. The geometric means and back-transformed 95% confidence intervals after a single dose of ridaforolimus and after multiple doses of ridaforolimus are presented for AUC0-24hr.
Time Frame: Cycle 1 Day 1: Predose and at various time points up to 24 hours postdose on Day 1; Cycle 1 Day 19: Predose and at various time points up to 24 hours postdose on Day 19; Cycle 1 is 19 days
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Ridaforolimus 40 mg
Number analyzed (Participants) | 13
ng*hr/mL
  Day 1 | 1846 [1361 to 2503]
  Day 19 | 2014 [1485 to 2731]

5. Primary Outcome: Maximum Concentration (Cmax) of Ridaforolimus: Day 1, Day 19
Description: Cmax is the peak blood plasma concentration following a dose of ridaforolimus. The (geometric) mean was calculated based on the back-transformed least-squares mean and the 95% confidence interval was determined from a linear mixed-effect model, containing a fixed effect for day and a random effect for participant, performed on natural log-transformed values. The geometric means and back-transformed 95% confidence intervals after a single dose of ridaforolimus and after multiple doses of ridaforolimus are presented for Cmax.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Ridaforolimus 40 mg
Number analyzed (Participants) | 13
ng/mL
  Day 1 | 210 [150 to 295]
  Day 19 | 167 [119 to 234]

6. Primary Outcome: Concentration at 24 Hours (C24hr) of Ridaforolimus: Day 1, Day 19
Description: C24hr is the concentration of ridaforolimus in the blood 24 hours after a dose of ridaforolimus. The (geometric) mean was calculated based on the back-transformed least-squares mean and the 95% confidence interval was determined from a linear mixed-effect model, containing a fixed effect for day and a random effect for participant, performed on natural log-transformed values. The geometric means and back-transformed 95% confidence intervals after a single dose of ridaforolimus and after multiple doses of ridaforolimus are presented for C24hr.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Ridaforolimus 40 mg
Number analyzed (Participants) | 15
ng/mL
  Day 1 | 34.8 [26.0 to 46.8]
  Day 19: number analyzed (Participants) | 13
  Day 19 | 49.7 [36.4 to 67.7]

7. Primary Outcome: Time to Maximum Concentration (Tmax) of Ridaforolimus: Day 1, Day 19
Description: Tmax is the time at which the Cmax of ridaforolimus is reached. The medians and ranges (minimum, maximum) for Tmax after a single dose of ridaforolimus and after multiple doses of ridaforolimus are presented.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Ridaforolimus 40 mg
Number analyzed (Participants) | 13
Hours
  Day 1 | 4.03 [2.00 to 7.97]
  Day 19 | 4.00 [0.00 to 6.00]

8. Primary Outcome: Apparent Terminal Half-life (t1/2) of Ridaforolimus: Cycle 1 (Cycle 1 is 19 Days)
Description: t½ is the time that it takes for the concentration of ridaforolimus in the body to decrease by half. The (harmonic) means and 95% confidence intervals for t1/2 after a single dose of ridaforolimus and after multiple doses of ridaforolimus are presented.
Time Frame: Cycle 1: Predose on Day 1 and at various time points through to 24 hours postdose on Day 19; Cycle 1 is 19 days
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | Ridaforolimus 40 mg
Number analyzed (Participants) | 15
Hours | 52.9 [40.2 to 65.6]

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after last dose (Up to 26 weeks)
Description: The Safety Population consisted of all participants who received at least one dose of study treatment.
Arm/Group | Ridaforolimus 40 mg
All-Cause Mortality (participants affected / at risk) | 3/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus 40 mg (N=15)
Disease progression (General disorders) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ridaforolimus 40 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 12 (15)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 6 (8)
Paronychia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 4 (4)
Blood cholesterol increased (Investigations) | 5 (6)
Gamma-glutamyltransferase increased (Investigations) | 6 (6)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 5 (9)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 8 (13)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.